CLINICAL TRIAL: NCT00091832
Title: A Randomized Active-controlled Study of AMG 162 in Breast Cancer Subjects With Bone Metastasis Who Have Not Previously Been Treated With Bisphosphonate Therapy.
Brief Title: Denosumab (AMG 162) in Bisphosphonate Naive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20040113
Record Dates: First submitted 2004-09-17; First posted 2004-09-21 (Estimated); Results first posted 2011-01-07 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer; Metastases; Bone Metastases in Subjects With Advanced Breast Cancer
Keywords: Breast Cancer; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Denosumab; Diphosphonates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Denosumab 60 mg every 12 weeks (Experimental): Denosumab 60 mg by subcutaneous injection once every 12 weeks (Q12W) for 25 weeks.
  Interventions: Biological: Denosumab
- Denosumab 120 mg every 4 weeks (Experimental): Denosumab 120 mg by subcutaneous injection once every 4 weeks (Q4W) for 25 weeks.
  Interventions: Biological: Denosumab
- Denosumab 180 mg every 4 weeks (Experimental): Denosumab 180 mg by subcutaneous injection once every 4 weeks (Q4W) for 25 weeks.
  Interventions: Biological: Denosumab
- IV bisphosphonates every 4 weeks (Active Comparator): Open label bisphosphonate every 4 weeks (Q4W) by intravenous infusion for 25 weeks.
  Interventions: Drug: IV Bisphosphonates
- Denosumab 180 mg every 12 weeks (Experimental): Denosumab 180 mg by subcutaneous injection once every 12 weeks (Q12W) for 25 weeks.
  Interventions: Biological: Denosumab
- Denosumab 30 mg every 4 weeks (Experimental): Denosumab 30 mg by subcutaneous injection once every 4 weeks (Q4W) for 25 weeks.
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — Denosumab administered by subcutaneous injection
  Other Names: AMG 162
  Arms: Denosumab 120 mg every 4 weeks; Denosumab 180 mg every 12 weeks; Denosumab 180 mg every 4 weeks; Denosumab 30 mg every 4 weeks; Denosumab 60 mg every 12 weeks
Drug: IV Bisphosphonates — Commercially available intravenous (IV) bisphosphonates administered per package insert, included pamidronate, ibandronic acid, and zoledronic acid
  Arms: IV bisphosphonates every 4 weeks

SUMMARY:
This study is to evaluate various doses and schedules for denosumab administration and characterize the safety profile in this indication.

ELIGIBILITY:
Inclusion Criteria: - Histologically or cytologically confirmed breast adenocarcinoma

* At least one bone metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2004-09; Primary Completion 2005-11 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Campbell-Baird C, Lipton A, Sarkenshik M, Ma H, Jun S.Incidence of Acute Phase Events Following Denosumab or Intravenous Bisphosphonates: Results From a Randomized, Controlled Phase 2 Study in Patients With Breast Cancer and Bone Metastases.Journal-001752;2010;7:85-89.
- [Background] Lipton A, Steger GG, Figueroa J, Alvarado C, Solal-Celigny P, Body JJ, de Boer R, Berardi R, Gascon P, Tonkin KS, Coleman RE, Paterson AH, Gao GM, Kinsey AC, Peterson MC, Jun S. Extended efficacy and safety of denosumab in breast cancer patients with bone metastases not receiving prior bisphosphonate therapy. Clin Cancer Res. 2008 Oct 15;14(20):6690-6. doi: 10.1158/1078-0432.CCR-07-5234. PMID 18927312
- [Background] Lipton A, Steger GG, Figueroa J, Alvarado C, Solal-Celigny P, Body JJ, de Boer R, Berardi R, Gascon P, Tonkin KS, Coleman R, Paterson AH, Peterson MC, Fan M, Kinsey A, Jun S. Randomized active-controlled phase II study of denosumab efficacy and safety in patients with breast cancer-related bone metastases. J Clin Oncol. 2007 Oct 1;25(28):4431-7. doi: 10.1200/JCO.2007.11.8604. Epub 2007 Sep 4. PMID 17785705
- [Background] Peterson M, Rodriquez R., Gurrola E., Sohn W, Jun S (others??).Population pharmacokinetics and pharmacodynamics of denosumab in breast cancer patients with bone metastases.Journal-000709;
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 8 September 2004 through 9 May 2005
Groups:
- Bisphosphonate IV Q4W: Open label bisphosphonate every 4 weeks (Q4W) by intravenous infusion (IV)
- Denosumab 30 mg Q4W: Denosumab 30 mg by subcutaneous injection every 4 weeks (Q4W)
- Denosumab 120 mg Q4W: Denosumab 120 mg by subcutaneous injection every 4 weeks (Q4W)
- Denosumab 180 mg Q4W: Denosumab 180 mg by subcutaneous injection every 4 weeks (Q4W)
- Denosumab 60 mg Q12W: Denosumab 60 mg by subcutaneous injection every 12 weeks (Q12W)
- Denosumab 180 mg Q12W: Denosumab 180 mg by subcutaneous injection every 12 weeks (Q12W)
Period: Overall Study
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Started | 43 | 42 | 42 | 43 | 42 | 43
Received Study Medication | 43 | 42 | 41 | 43 | 42 | 43
Completed | 29 | 31 | 30 | 29 | 27 | 32
Not Completed | 14 | 11 | 12 | 14 | 15 | 11
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 0 | 1 | 3 | 1
Not completed — Death | 6 | 4 | 5 | 8 | 5 | 6
Not completed — Disease Progression | 2 | 0 | 0 | 1 | 1 | 2
Not completed — Ineligibility Determined | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 3 | 3 | 2 | 1
Not completed — Noncompliance | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bisphosphonate IV Q4W: Open label bisphosphonate every 4 weeks (Q4W) by intravenous infusion
- Total: Total of all reporting groups
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Total
Number analyzed (Participants) | 43 | 42 | 42 | 43 | 42 | 43 | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (10.7) | 56.5 (10.8) | 59.2 (12.3) | 58.2 (9.1) | 57.4 (11.0) | 57.6 (13.9) | 57.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 42 | 43 | 42 | 43 | 255
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 25 | 28 | 29 | 34 | 30 | 33 | 179
  Hispanic or Latino | 16 | 13 | 13 | 9 | 10 | 10 | 71
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Other | 1 | 0 | 0 | 0 | 1 | 0 | 2
uNTx/Cr [Mean (Standard Deviation); unit: nmol/mmol] — Urinary N-telopeptide corrected by creatinine (uNTx/Cr)
  nmol/mmol | 83.16 (94.37) | 66.44 (61.17) | 89.41 (98.58) | 75.92 (91.03) | 102.06 (129.12) | 98.22 (168.42) | 85.78 (111.94)
Serum CTx [Mean (Standard Deviation); unit: ng/mL] — Type I serum C-Telopeptide (CTx)
  ng/mL | 0.592 (0.284) | 0.632 (0.430) | 0.720 (0.559) | 0.647 (0.703) | 0.714 (0.564) | 0.846 (0.892) | 0.692 (0.605)
TRAP 5b [Mean (Standard Deviation); unit: U/L] — Tartrate-resistant acid phosphatase 5b (TRAP 5b)
  U/L | 6.907 (3.280) | 6.879 (2.878) | 7.116 (3.493) | 7.628 (6.830) | 6.765 (4.340) | 7.009 (4.217) | 7.057 (4.358)
BSAP [Mean (Standard Deviation); unit: U/L] — Bone specific alkaline phosphatase (BSAP)
  U/L | 54.84 (51.69) | 44.33 (26.06) | 45.62 (26.02) | 62.39 (109.18) | 47.89 (30.46) | 48.82 (35.13) | 50.75 (55.04)
P1NP [Mean (Standard Deviation); unit: µg/L] — Procollagen 1 N-terminal peptide (P1NP)
  µg/L | 111.01 (97.21) | 98.54 (72.69) | 114.29 (113.51) | 193.03 (641.13) | 98.47 (83.46) | 139.01 (188.02) | 126.20 (284.81)
Osleocalcin [Mean (Standard Deviation); unit: ng/mL] | 9.42 (5.89) | 9.25 (4.98) | 10.04 (5.70) | 8.96 (5.03) | 8.09 (3.36) | 9.31 (4.06) | 9.20 (4.93)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 13 in Creatinine-adjusted Urinary N-telopeptide (uNTx/Cr)
Description: Percent change from Baseline to Week 13 in Urinary N-telopeptide corrected by creatinine (uNTx/Cr) calculated using ((Week 13 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and Week 13
Population: Primary Efficacy Subset, composed of all participants who were randomized, received at least one dose of denosumab or bisphosphonate, and had both a baseline and at least one postbaseline measurement of Urinary N-telopeptide corrected by creatinine (uNTx/Cr). Analysis was by Intention-to-Treat (ITT).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 38 | 40 | 38 | 40 | 38 | 40
Percent change | -10.19 (208.84) | -52.87 (95.14) | -54.21 (61.34) | -57.36 (41.46) | -51.73 (60.85) | -18.46 (125.86)
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 30 mg Q4W vs Denosumab 120 mg Q4W vs Denosumab 180 mg Q4W vs Denosumab 60 mg Q12W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; p = 0.245, ANCOVA; Adjusted for the stratum to which the participant was originally assigned by the Interactive Voice Response System (IVRS)

2. Secondary Outcome: Percent Change From Baseline to Week 25 in Urinary N-telopeptide (uNTx)
Description: Percent change from Baseline to Week 25 in Urinary N-telopeptide (uNTx) calculated using ((Week 25 value - Baseline value) / Baseline value) x 100.
Time Frame: Baseline and Week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 34 | 36 | 34 | 38 | 32 | 35
Percent change | -39.52 (74.16) | -53.46 (100.77) | -43.16 (101.08) | -59.41 (43.31) | -41.79 (72.61) | -39.96 (65.85)
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 30 mg Q4W vs Denosumab 120 mg Q4W vs Denosumab 180 mg Q4W vs Denosumab 60 mg Q12W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; p = 0.848, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants Achieving 65% or More Reduction in Urinary N-telopeptide (uNTx) From Baseline at Week 13
Description: The number of participants achieving a 65% reduction or more in uNTx from Baseline at Week 13. Calculation used is ((Week 13 value - Baseline value) / Baseline value ) x 100 and participants were considered having a 65% reduction or more if their value was ≤ -65%.
Time Frame: Baseline and Week 13
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 41 | 41 | 40 | 43 | 42 | 42
Participants | 25 | 24 | 26 | 24 | 20 | 21
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 60 mg Q12W; Test type: Superiority or Other; Odds Ratio (OR) = 1.72, 95% CI [0.68 to 4.35] — Adjusted for the stratum to which the participant was originally assigned by the Interactive Voice Response System (IVRS)
Statistical Analysis 2: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; Odds Ratio (OR) = 1.29, 95% CI [0.51 to 3.24] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Bisphosphonate IV Q4W vs Denosumab 120 mg Q4W; Test type: Superiority or Other; Odds Ratio (OR) = 0.88, 95% CI [0.34 to 2.29] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Bisphosphonate IV Q4W vs Denosumab 30 mg Q4W; Test type: Superiority or Other; Odds Ratio (OR) = 1.27, 95% CI [0.51 to 3.20] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; Odds Ratio (OR) = 1.74, 95% CI [0.70 to 4.34] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Number of Participants Achieving 65% or More Reduction in uNTX From Baseline at Week 25
Description: The number of participants achieving a 65% reduction or more in uNTX from Baseline at Week 25. Calculation used is ((Week 25 value - Baseline value) / Baseline value) x 100 and participants were considered having a 65% reduction or more if their value was ≤ -65%.
Time Frame: Baseline and Week 25
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 41 | 41 | 40 | 43 | 42 | 42
Participants | 19 | 25 | 23 | 25 | 21 | 15
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; Odds Ratio (OR) = 1.82, 95% CI [0.69 to 4.79] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; Odds Ratio (OR) = 0.67, 95% CI [0.25 to 1.76] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Bisphosphonate IV Q4W vs Denosumab 120 mg Q4W; Test type: Superiority or Other; Odds Ratio (OR) = 0.65, 95% CI [0.24 to 1.77] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Bisphosphonate IV Q4W vs Denosumab 30 mg Q4W; Test type: Superiority or Other; Odds Ratio (OR) = 0.58, 95% CI [0.22 to 1.58] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Bisphosphonate IV Q4W vs Denosumab 60 mg Q12W; Test type: Superiority or Other; Odds Ratio (OR) = 0.70, 95% CI [0.25 to 1.92] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Time to 65% or More Reduction in Urinary N-telopeptide (uNTX) From Baseline
Description: Kaplan-Meier estimate of the median time from enrollment to the first occurrence of a reduction of uNTx of ≥ 65% compared to Baseline. For participants whose uNTx did not fall below 65% of the Baseline value, the time was censored at time of last evaluation of uNTx.
Time Frame: Baseline to Week 57
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 41 | 41 | 40 | 43 | 42 | 42
Days | 10 [8 to 86] | 13 [8 to 57] | 11 [9 to 43] | 10 [8 to 42] | 9 [8 to 29] | 30 [9 to 141]
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; Hazard Ratio (HR) = 0.82, 95% CI [0.51 to 1.31] — A hazard ratio >1 indicates that the time to 65% or more reduction in uNTx from baseline was shorter in the Denosumab-treated group than in the control group
Statistical Analysis 2: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; Hazard Ratio (HR) = 1.03, 95% CI [0.64 to 1.65] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Bisphosphonate IV Q4W vs Denosumab 120 mg Q4W; Test type: Superiority or Other; Hazard Ratio (HR) = 1.09, 95% CI [0.68 to 1.74] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Bisphosphonate IV Q4W vs Denosumab 30 mg Q4W; Test type: Superiority or Other; Hazard Ratio (HR) = 1.09, 95% CI [0.68 to 1.74] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Bisphosphonate IV Q4W vs Denosumab 60 mg Q12W; Test type: Superiority or Other; Hazard Ratio (HR) = 1.14, 95% CI [0.71 to 1.83] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percent Change From Baseline to Week 13 in Serum C-Telopeptide (CTX)
Description: Percent change from Baseline to Week 13 in type I serum C-telopeptide (CTX) calculated using ((Week 13 value - Baseline value) / Baseline value) x 100.
Time Frame: Baseline and week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 38 | 39 | 38 | 40 | 38 | 40
Percent change | -66.92 (44.05) | -80.76 (12.66) | -78.45 (28.89) | -81.79 (13.29) | -70.50 (41.76) | -78.13 (16.66)

7. Secondary Outcome: Percent Change From Baseline to Week 25 in Serum C-telopeptide (CTX)
Description: Percent change from Baseline to Week 25 in type I serum C-telopeptide calculated using ((Week 25 value - Baseline value) / Baseline value) x 100.
Time Frame: Baseline and Week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 34 | 36 | 34 | 38 | 33 | 35
Percent change | -73.09 (22.42) | -82.70 (11.92) | -74.48 (30.26) | -80.07 (22.26) | -70.64 (36.94) | -78.31 (14.00)

8. Secondary Outcome: Percent Change From Baseline to Week 13 in Procollagen I N-terminal Peptide (P1NP)
Description: Percent change from Baseline to Week 13 in procollagen 1 N-terminal peptide calculated using ((Week 13 value - Baseline value) / Baseline value) x 100.
Time Frame: Baseline and Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 37 | 39 | 37 | 40 | 38 | 40
Percent change | -50.75 (29.47) | -52.35 (36.90) | -48.23 (36.83) | -50.47 (54.67) | -43.94 (44.53) | -59.42 (18.60)

9. Secondary Outcome: Percent Change From Baseline to Week 25 in P1NP
Description: Percent change from Baseline to Week 25 in procollagen 1 N-terminal peptide (P1NP) calculated using ((Week 25 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and Week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 34 | 36 | 34 | 37 | 33 | 35
Percent change | -50.48 (41.22) | -53.48 (54.79) | -55.90 (30.66) | -57.88 (51.97) | -51.18 (40.41) | -51.37 (47.53)

10. Secondary Outcome: Percent Change From Baseline to Week 13 in Tartrate-resistant Acid Phosphatase 5b (TRAP5b)
Description: Percent change from Baseline to Week 13 in tartrate-resistant acid phosphatase 5b calculated using ((Week 13 value - Baseline value) / Baseline value) x 100.
Time Frame: Baseline and Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 36 | 38 | 35 | 37 | 35 | 39
Percent change | -37.45 (19.87) | -56.07 (17.80) | -58.24 (15.07) | -53.12 (50.00) | -55.85 (27.22) | -55.91 (17.61)

11. Secondary Outcome: Percent Change From Baseline to Week 25 in Tartrate-resistant Acid Phosphatase 5b (TRAP5b)
Description: Percent change from Baseline to Week 25 in TRAP5b calculated using ((Week 25 value - Baseline value) / Baseline value) x 100.
Time Frame: Baseline and Week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 33 | 35 | 32 | 35 | 30 | 33
Percent change | -38.59 (26.06) | -58.58 (18.93) | -52.39 (25.30) | -51.15 (44.49) | -56.25 (32.30) | -53.13 (22.23)

12. Secondary Outcome: Percent Change From Baseline to Week 13 in Bone Specific Alkaline Phosphatase (BSAP)
Description: Percent change from Baseline to Week 13 in bone specific alkaline phosphatase (BSAP) calculated using ((Week 13 value - Baseline value) / Baseline value) x 100.
Time Frame: Baseline and Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 36 | 38 | 35 | 39 | 37 | 38
Percent change | -40.01 (24.42) | 26.37 (406.79) | -40.23 (27.34) | -38.42 (25.44) | -37.11 (31.33) | -35.94 (25.49)

13. Secondary Outcome: Percent Change From Baseline to Week 25 in Bone Specific Alkaline Phosphatase (BSAP)
Description: Percent change from Baseline to Week 25 in BSAP calculated using ((Week 25 value - Baseline value) / Baseline value) x 100.
Time Frame: Baseline and Week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 34 | 35 | 32 | 35 | 32 | 33
Percent change | -46.56 (26.02) | 15.88 (347.47) | -49.01 (21.24) | -52.60 (16.23) | -46.72 (23.25) | -48.24 (27.61)

14. Secondary Outcome: Percent Change From Baseline to Week 13 in Osteocalcin
Description: Percent change from Baseline to Week 13 in osteocalcin calculated using ((Week 13 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 36 | 38 | 35 | 39 | 37 | 38
Percent change | 6.82 (49.78) | -19.35 (38.71) | -2.39 (47.96) | -6.23 (40.82) | -23.78 (35.46) | -5.96 (41.92)

15. Secondary Outcome: Percent Change From Baseline to Week 25 in Osteocalcin
Description: Percent change from Baseline to Week 25 in osteocalcin calculated using ((Week 25 value - Baseline value) / Baseline value) x 100.
Time Frame: Baseline and Week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 34 | 35 | 32 | 35 | 32 | 33
Percent change | -4.74 (86.98) | -30.78 (34.94) | -22.80 (46.36) | -26.95 (41.49) | -23.93 (43.99) | -22.69 (36.79)

16. Secondary Outcome: Time to First Skeletal Related Event
Description: Skeletal Related Event (SRE) defined as ≥ 1 of the following: pathological bone fracture, spinal cord compression, surgery or radiation therapy to bone (including the use of radioisotopes).
Time Frame: Day 1 to Week 25
Population: All participants who were exposed to investigational product.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 43 | 42 | 41 | 43 | 42 | 43
Days | NA [NA to NA] — Median could not be calculated due to the low number of skeletal-related events | NA [NA to NA] — Median could not be calculated due to the low number of skeletal-related events | NA [NA to NA] — Median could not be calculated due to the low number of skeletal-related events | NA [NA to NA] — Median could not be calculated due to the low number of skeletal-related events | NA [NA to NA] — Median could not be calculated due to the low number of skeletal-related events | NA [NA to NA] — Median could not be calculated due to the low number of skeletal-related events
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 30 mg Q4W; Test type: Superiority or Other; Hazard Ratio (HR) = 0.543, 95% CI [0.159 to 1.856] — A hazard ratio <1 indicates the time to the first skeletal-related event in the denosumab-treated group was longer than that in the control group
Statistical Analysis 2: Comparison: Bisphosphonate IV Q4W vs Denosumab 60 mg Q12W; Test type: Superiority or Other; Hazard Ratio (HR) = 0.544, 95% CI [0.159 to 1.859] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 3: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; Hazard Ratio (HR) = 0.791, 95% CI [0.266 to 2.355] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 4: Comparison: Bisphosphonate IV Q4W vs Denosumab 120 mg Q4W; Test type: Superiority or Other; Hazard Ratio (HR) = 1.073, 95% CI [0.389 to 2.963] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 5: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; Hazard Ratio (HR) = 0.540, 95% CI [0.158 to 1.847] — [estimate comment as in outcome 16, analysis 1]

17. Secondary Outcome: Number of Participants With Skeletal Related Events
Description: Skeletal Related Events (SRE) are defined as ≥ 1 of the following: pathological bone fracture, spinal cord compression, surgery or radiation therapy to bone (including the use of radioisotopes).
Time Frame: From Day 1 to Week 25
Population: All participants who were exposed to investigational product.
Measure: Number; unit: Participants
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 43 | 42 | 41 | 43 | 42 | 43
Participants | 7 | 4 | 8 | 6 | 4 | 4
Statistical Analysis 1: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q12W; Test type: Superiority or Other; Odds Ratio (OR) = 1.92, 95% CI [0.51 to 7.17] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Bisphosphonate IV Q4W vs Denosumab 180 mg Q4W; Test type: Superiority or Other; Odds Ratio (OR) = 1.20, 95% CI [0.36 to 3.97] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Bisphosphonate IV Q4W vs Denosumab 120 mg Q4W; Test type: Superiority or Other; Odds Ratio (OR) = 0.81, 95% CI [0.26 to 2.52] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Bisphosphonate IV Q4W vs Denosumab 60 mg Q12W; Test type: Superiority or Other; Odds Ratio (OR) = 1.88, 95% CI [0.5 to 7.05] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Bisphosphonate IV Q4W vs Denosumab 30 mg Q4W; Test type: Superiority or Other; Odds Ratio (OR) = 1.88, 95% CI [0.5 to 7.05] — [estimate comment as in outcome 3, analysis 1]

18. Secondary Outcome: Number of Participants With Hypercalcemia
Description: Occurrence of grade 3 or 4 hypercalcemia according to the Common Terminology Criteria for Adverse Events (CTCAE) v3. A summary of hypercalcemia events is reported under adverse events.
Time Frame: Day 1 to Week 57
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Number analyzed (Participants) | 41 | 41 | 40 | 43 | 42 | 42
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 25 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Bisphosphonate IV Q4W | Denosumab 30 mg Q4W | Denosumab 120 mg Q4W | Denosumab 180 mg Q4W | Denosumab 60 mg Q12W | Denosumab 180 mg Q12W
Serious Adverse Events (participants affected / at risk) | 15/43 | 11/42 | 19/41 | 16/43 | 14/42 | 15/43
Other Adverse Events (participants affected / at risk) | 36/43 | 33/42 | 37/41 | 36/43 | 37/42 | 35/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisphosphonate IV Q4W (N=43) | Denosumab 30 mg Q4W (N=42) | Denosumab 120 mg Q4W (N=41) | Denosumab 180 mg Q4W (N=43) | Denosumab 60 mg Q12W (N=42) | Denosumab 180 mg Q12W (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 0 | 2 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 4 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 1 | 0 | 0 | 1 | 1
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Central line infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Neurocysticercosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Karnofsky scale worsened (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 0 | 0
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0 | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Internal fixation of fracture (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Secondary hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bisphosphonate IV Q4W (N=43) | Denosumab 30 mg Q4W (N=42) | Denosumab 120 mg Q4W (N=41) | Denosumab 180 mg Q4W (N=43) | Denosumab 60 mg Q12W (N=42) | Denosumab 180 mg Q12W (N=43)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 2 | 7 | 5
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 2 | 3 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 3 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 1 | 4 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 0 | 1 | 3 | 1
Constipation (Gastrointestinal disorders) | 7 | 7 | 5 | 6 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 9 | 9 | 6 | 4 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 3 | 1
Nausea (Gastrointestinal disorders) | 10 | 10 | 9 | 11 | 7 | 9
Vomiting (Gastrointestinal disorders) | 8 | 11 | 7 | 5 | 7 | 4
Asthenia (General disorders) | 12 | 9 | 9 | 4 | 6 | 5
Fatigue (General disorders) | 5 | 7 | 5 | 5 | 6 | 5
Injection site pain (General disorders) | 0 | 0 | 1 | 3 | 1 | 0
Mucosal inflammation (General disorders) | 1 | 3 | 0 | 1 | 3 | 1
Oedema peripheral (General disorders) | 5 | 2 | 0 | 3 | 2 | 6
Pain (General disorders) | 2 | 3 | 0 | 3 | 3 | 2
Pyrexia (General disorders) | 8 | 2 | 4 | 3 | 3 | 3
Influenza (Infections and infestations) | 3 | 1 | 0 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 2 | 1 | 5
Anorexia (Metabolism and nutrition disorders) | 3 | 6 | 3 | 5 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 3 | 4 | 9 | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 9 | 5 | 4 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 2 | 7 | 6 | 5 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 3 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 3 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 3 | 1 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 6 | 4 | 6 | 2 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 2 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 0 | 3 | 1
Headache (Nervous system disorders) | 7 | 4 | 6 | 6 | 8 | 4
Lethargy (Nervous system disorders) | 2 | 1 | 4 | 1 | 1 | 1
Neuralgia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 4 | 1 | 3 | 3 | 3 | 1
Depression (Psychiatric disorders) | 3 | 2 | 2 | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 3 | 1 | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 5 | 2 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3 | 3 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 3 | 3 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 2 | 1 | 3
Radiotherapy to bone (Surgical and medical procedures) | 3 | 2 | 3 | 2 | 2 | 1
Hot flush (Vascular disorders) | 2 | 3 | 5 | 0 | 2 | 2
Hypertension (Vascular disorders) | 3 | 2 | 0 | 2 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.